CLINICAL TRIAL: NCT03483298
Title: Prospective Split Cohort Trial Comparing in Vitro Fertilization (IVF) Outcomes After the Use of Testicular Versus Ejaculated Sperm for ICSI in Med With Elevated DNA Fragmentation After a Failed IVF Cycle
Brief Title: Split Cohort Trial Comparing IVF Outcomes After the Use of Testicular vs. Ejaculated Sperm for ICSI
Status: Terminated | Type: Observational
Why Stopped: recruitment issues
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-2018-04
Record Dates: First submitted 2018-03-23; First posted 2018-03-30 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum obtained from male patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- elevated sperm DNA fragmentation: Couples with male partners who will be undergoing a TESA procedure secondary to elevated DNA fragmentation (>25% DFI) as part of their routine IVF treatment will have half of the women's eggs inseminated with ejaculated sperm and the other half with surgically obtained sperm via the ICSI procedure
  Interventions: Other: ICSI

INTERVENTIONS:
Other: ICSI — The cryopreserved pre-TESA ejaculate and TESA specimen will be thawed on the day of oocyte retrieval per protocol for ICSI

SUMMARY:
The primary objective of this study is to determine if there is a difference in in vitro fertilization (IVF) with intracytoplasmic sperm injection (ICSI) outcomes when using testicular sperm versus ejaculated sperm in couples with elevated sperm DNA fragmentation after a failed in vitro fertilization (IVF) cycle

DETAILED DESCRIPTION:
The experimental design for this study is as follows:

1. Couples with male partners who will be undergoing a TESA procedure secondary to elevated DNA fragmentation (>25% DFI) as part of their routine IVF treatment will be contacted for possible study participation.
2. Informed consent will be obtained
3. The primary investigator will be notified of the couple's participation.
4. The male partner will cryopreserve an ejaculated semen sample if there is no cryopreserved ejaculated specimen in inventory. The male partner will undergo a surgical sperm retrieval (TESA) and the specimen will be frozen per routine.
5. Serum will be collected from the male partner and preserved for future analysis.
6. The cryopreserved pre-TESA ejaculate and TESA specimen will be thawed on the day of oocyte retrieval per protocol. After oocyte retrieval, oocytes will be analyzed per routine and assessed for maturity. The oocytes will be divided into two groups per embryologist discretion. One group will be labeled 'A' and the other will be labeled B.' A random letter generator will create a list of 'A' and 'B's which will be placed in sequentially numbered, sealed envelopes. The envelopes will be opened in sequence according to patient enrollment. The first envelope opened by the embryologist will reveal the letter of the oocyte group that will be inseminated with testicular sperm. The other group will be inseminated with the frozen/ thawed ejaculated sperm. Therefore, half of the oocytes will be inseminated using intracytoplasmic sperm injection (ICSI) with testicular sperm and the other half will be inseminated via ICSI with ejaculated sperm. If there are an odd number of oocytes, the extra oocyte will always belong to group A for simplicity.
7. If fertilized, the group of zygotes created using testicular sperm will take the group letter that corresponded to the testicular sperm. This will also be true of the zygotes using ejaculated sperm. Both groups of zygotes will be cultured to the blastocyst stage with culture conditions per standard laboratory procedures.
8. Fertilization and blastulation rates of the two groups will be recorded for each patient.
9. Each blastocyst will be biopsied for comprehensive chromosome screening (CCS) in routine fashion. Once comprehensive chromosomal screening results are available, if at least one euploid embryo is available, patients will undergo a single embryo transfer in a subsequent menstrual cycle.
10. Frozen embryo transfer cycles will be performed using either a programmed cycle (exogenous estradiol with subsequent progesterone) or a natural cycle to prepare the endometrium for embryo transfer.
11. If at least one euploid embryo is available from each group, a second randomization will occur at the time of embryo selection. The embryologist selecting the embryo for transfer will open a second sealed envelope, which contains the letter of the group from which the embryo for transfer should reside. The best quality embryo (per embryologist discretion) from the group corresponding to the letter in this envelope will be selected for transfer. The embryologist selecting the embryo will be blinded as to which group of embryos was created with ejaculated versus testicular sperm. The group from which the embryo selected for transfer was derived will be recorded.
12. Both the patient and the physician performing the embryo transfer will be blinded with regard to the group from which the embryo selected for transfer derived.
13. Pregnancy testing and follow up will proceed as per routine.
14. Approximately 8 weeks post-transfer, each participant will be assigned a cycle outcome (i.e., no pregnancy, miscarriage, ongoing pregnancy). At that time, the study participants can be notified of whether the sperm utilized for ICSI was derived from testicular sperm or ejaculated sperm. This information could be shared via telephone or in-person.

ELIGIBILITY:
Inclusion Criteria:

* Willing to comply with all study procedures and be available for the duration of the study
* Failed at least one IVF cycle (i.e., no live birth)
* Elevated DNA fragmentation noted in ejaculated sperm (>25% DFI according to the American Society of Reproductive Medicine guidelines)
* Couple electing single embryo transfer
* Couples electing comprehensive chromosome screening (CCS) of embryos
* At least 4 oocytes retrieved in IVF cycle in order to randomize

Exclusion Criteria:

* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.
* Contraindication to IVF
* Clinical indication for preimplantation genetic diagnosis (PGD) (i.e., screening for single gene disorder, chromosomal translocation, or any other disorders requiring detailed embryo genetic analysis)
* Male partner with azoospermia (<100,000 motile spermatozoa)
* Male partner with Y-chromosome microdeletion
* Male partner with any Karyotype other than 46,XY(normal male karyotype)
* Female partner history of hydrosalpinges or adnexal mass
* Female partner history of endometrial insufficiency (max endometrial thickness < 7mm)
* Female partner BMI < 35

Ages: 18 Years to 65 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Men with Elevated DNA fragmentation noted in ejaculated sperm (>25% DFI according to the American Society of Reproductive Medicine guidelines) and one prior failed IVF cycle
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-06-23 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Blastulation Rate of testicular vs. ejaculated sperm after ICSI | 1 week post ICSI
  # blast per 2 pronuclei in each group

SECONDARY OUTCOMES:
Fertilization Rate | 24 hrs post ICSI
  # fertilized per M2 in each group
Aneuploidy Rate | approximately 2 weeks post trophectoderm biopsy
  # abnormal embryos per useable blast in each group
Clinical Pregnancy Rate | approximately 2 weeks post pregnancy test
  defined by presence of gestational sac and yolk sac in uterus on ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Phil Cheng, MD, Principal Investigator — IVI RMA
Locations (1):
- IVI RMA New Jersey, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Esteves SC, Sanchez-Martin F, Sanchez-Martin P, Schneider DT, Gosalvez J. Comparison of reproductive outcome in oligozoospermic men with high sperm DNA fragmentation undergoing intracytoplasmic sperm injection with ejaculated and testicular sperm. Fertil Steril. 2015 Dec;104(6):1398-405. doi: 10.1016/j.fertnstert.2015.08.028. Epub 2015 Oct 1. PMID 26428305
- [Background] Greco E, Scarselli F, Iacobelli M, Rienzi L, Ubaldi F, Ferrero S, Franco G, Anniballo N, Mendoza C, Tesarik J. Efficient treatment of infertility due to sperm DNA damage by ICSI with testicular spermatozoa. Hum Reprod. 2005 Jan;20(1):226-30. doi: 10.1093/humrep/deh590. Epub 2004 Nov 11. PMID 15539441
- [Background] Bradley CK, McArthur SJ, Gee AJ, Weiss KA, Schmidt U, Toogood L. Intervention improves assisted conception intracytoplasmic sperm injection outcomes for patients with high levels of sperm DNA fragmentation: a retrospective analysis. Andrology. 2016 Sep;4(5):903-10. doi: 10.1111/andr.12215. Epub 2016 May 27. PMID 27231097
- [Background] Pabuccu EG, Caglar GS, Tangal S, Haliloglu AH, Pabuccu R. Testicular versus ejaculated spermatozoa in ICSI cycles of normozoospermic men with high sperm DNA fragmentation and previous ART failures. Andrologia. 2017 Mar;49(2). doi: 10.1111/and.12609. Epub 2016 Apr 25. PMID 27108915
- [Background] Mehta A, Bolyakov A, Schlegel PN, Paduch DA. Higher pregnancy rates using testicular sperm in men with severe oligospermia. Fertil Steril. 2015 Dec;104(6):1382-7. doi: 10.1016/j.fertnstert.2015.08.008. Epub 2015 Sep 9. PMID 26363389
- [Background] Lewis SE, John Aitken R, Conner SJ, Iuliis GD, Evenson DP, Henkel R, Giwercman A, Gharagozloo P. The impact of sperm DNA damage in assisted conception and beyond: recent advances in diagnosis and treatment. Reprod Biomed Online. 2013 Oct;27(4):325-37. doi: 10.1016/j.rbmo.2013.06.014. Epub 2013 Jul 11. PMID 23948450